CLINICAL TRIAL: NCT05813704
Title: A Prospective, Multicenter Clinical Trial in Evaluating the Safety and Efficacy of the Coronary Crossing System in Patients With Coronary Chronic Total Occlusions
Brief Title: Coronary Crossing System in Patients With Coronary Chronic Total Occlusions
Acronym: VITAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Shanghai Baoshan District Wusong Central Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Tianjin First Central Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Hebei General Hospital (Other); West China Hospital (Other); First Affiliated Hospital of Army Medical University, PLA (Unknown); Lanzhou University First Hospital (Unknown); Nanfang Hospital, Southern Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD-D-003
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: chronic total occlusions; coronary artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary Crossing System (Experimental): Subjects in experimental group will be treated with the Coronary Crossing System manufactured by Shanghai Microport Rhythm Co. Ltd.
  Interventions: Device: Coronary Crossing System of Shanghai MicroPort Rhythm

INTERVENTIONS:
Device: Coronary Crossing System of Shanghai MicroPort Rhythm — The mechanical vibration generated by the Coronary Crossing System through the piezoelectric effect is amplified and transmitted to the distal end of the guidewire to achieve high-frequency vibration at the tip of the guidewire, and then achieve efficient and safe penetration of the fibrous cap of the CTO.

SUMMARY:
This is a prospective and multicenter clinical investigation aiming to evaluate the safety and effectiveness of coronary crossing system for the treatment of patients with coronary chronic total occlusions.

DETAILED DESCRIPTION:
This study is divided into two phases. The first phase is the pilot study stage, which is a prospective single-group observational test (FIM phase). The second phase is the pivotal study phase, which is a prospective, multi-center, single-group clinical trial (OPC phase). It is carried out in about 20 hospitals in China.

1. Pilot study phase (FIM phase): It is a prospective single-group observational test. It is expected to recruit 10 subjects in a research center in China.
2. Pivotal study phase (OPC phase): It is a prospective, multicenter, single-group clinical trial. 146 subjects are expected to be recruited in 20 research centers in China.
3. All subjects with coronary chronic total occlusions participating in this clinical study must have only a CTO lesion which occluded in length of more than 5 mm and located in a native coronary artery with a diameter of ≥ 2.50 mm (visual inspection).
4. All subjects receive clinical follow-up during hospitalization, 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion Criteria:

1. Aged 18 years and older.
2. Subjects with coronary artery disease who have symptoms of angina pectoris and evidence of ischemia or myocardial viability in the area innervated by the coronary arteries where the CTO is located.
3. Subjects who are able to understand the purpose of the trial, participate voluntarily or by proxy and indicate by signing the informed consent form that they recognize the risks and benefits described in the informed consent document and are willing to undergo clinical follow-up.

Angiography Inclusion Criteria:

1. There is only one target CTO that needs to be treated with percutaneous coronary intervention (PCI).
2. Target CTO is located in a native coronary artery with a reference vessel diameter of ≥ 2.5 mm.
3. Angiography showed complete occlusion of the target CTO (visual inspection), antegrade flow of the occluded vessel segment TIMI grade 0 and inferred occlusion time ≥ 3 months; or previous angiographic records confirmed occluded time of the target CTO ≥ 3 months.
4. The target CTO occluded segment length ≥ 5 mm (visual inspection).
5. Angiography of the target CTO showed high density along the vessel, which is considered calcified lesion.
6. The antegrade approach is determined as the primary strategy with guidewire crossing in PCI treatment.
7. The fibrous cap of the target lesion can not be penetrated within 60 seconds using the guidewire with polypolymer coated or tip stiffness > 1.5g (visual inspection) under fluoroscopy and the time is timed when the guidewire reaches the fibrous cap. (To identify chronic total occlusions and exclude acute or subacute occlusions that such guidewire can pass directly).
8. In addition to the target lesion, there must be up to one non-target lesion to be treated and it is located on a different epicardial vessel than the target lesion. Target lesions can be treated after successful treatment of the non-target lesion (residual stenosis < 30% and TIMI 3 flow) without complications.

Exclusion Criteria:

General Exclusion Criteria:

1. Acute myocardial infarction within 30 days prior to baseline procedure.
2. Life expectancy < 1 year.
3. Inability to use protocol-required concomitant medications (eg, aspirin, P2Y12 platelet receptor inhibitors, heparin, contrast agents, etc) due to allergy or other contraindications, and no alternative medications.
4. The target CTO has an iatrogenic dissection that occurred within the past 3 months.
5. Left ventricular ejection fraction less than 35%.
6. Severe aortic or mitral valve disease.
7. Planned left ventricular (LV) support device during CTO PCI.
8. Subjects with clear bleeding tendency, contraindications to antiplatelet agents and anticoagulant therapy.
9. Stroke, transient ischemic attack (TIA), or significant gastrointestinal (GI) bleeding within 6 months before the baseline procedure.
10. Planned additional coronary or valvular percutaneous or surgical intervention scheduled within 30 days after baseline procedure.
11. Subjects who require emergent or urgent PCI.
12. Female subjects who are pregnant or breast-feeding.
13. Subjects who are participating in another investigational drug or device clinical trial in which the primary endpoint is still not reached, or intend to participate in another investigational drug or device clinical trial within 12 months after baseline procedure.
14. Other medical illnesses that may cause the subject to be non-compliant with the protocol or confound data interpretation.
15. Serum creatinine > 2.5 mg/dL (or 221 µmol/L), or on dialysis.
16. Hemodynamic instability or severely impaired activity tolerance (KILLIP Class III, IV, or NYHA Class III, IV).
17. Subjects with sustained tachyarrhythmia or cardiogenic shock.

Angiography Exclusion Criteria:

1. The target CTO is in an unprotected left main.
2. No angiographically visible collateral flow to the target vessel distal to the occlusion, from ipsilateral or contralateral collaterals.
3. Because of the presence of moderate to severe tortuosity or stenosis in the collateral vessels, retrograde approach is not preferred at the investigator 's discretion.
4. Vessel tortuosity proximal to, or within, body of target occlusion which, in the opinion of the investigator, is not amenable to advancement of a microcatheter or Coronary Crossing System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Device success | Baseline procedure
  Device success is defined as successful antegrade crossing of the CTO into the true arterial lumen distal to the occlusion following advancement of at least 3 mm of the Coronary Crossing System into any segment as assessed by the core angiographic laboratory.
  (An antegrade only approach may involve Antegrade Dissection Re-Entry (ADR) with or without the use of specialized devices (e.g. Stingray); absence of successful retrograde crossing of a collateral will still be considered an antegrade only approach.)

SECONDARY OUTCOMES:
Overall device success | Baseline procedure
  Overall device success is defined as successful crossing of the CTO, following use of the coronary crossing system during the procedure including antegrade or retrograde approach.
Technical Success | Baseline procedure
  Technical success is defined as successful antegrade or retrograde crossing of the CTO into the true arterial lumen following advancement of at least 3 mm of the Coronary Crossing System into the proximal segment, with <30% residual stenosis of the CTO after successful treatment with drug-eluting stents or drug-eluting balloons, with antegrade flow≥TIMI grade 2 in all branch vessels ≥ 2.5 mm in diameter distal to the CTO, as assessed by the core angiographic laboratory.
Procedural Success | Baseline procedure
  Procedural success is defined as the achievement of Technical Success with freedom from device related MAEs as assessed by the Clinical Events Committee (CEC).
Clinical Success | 30 days post-procedure
  Clinical success is defined as the achievement of Procedural Success with freedom from device related MAEs through 48 hours or hospital discharge and 30 days post index procedure as assessed by the Clinical Events Committee (CEC).
Freedom from device related major adverse event(MAE) | 48 hours or until discharge
  Freedom from device related major adverse events (MAEs) at 48 hours or hospital discharge (whichever occurs first) post procedure, as assessed by Clinical Events Committee (CEC), defined as:
  * Cardiovascular related deaths
  * Myocardial Infarction.
  * Coronary Artery Perforation requiring treatment
  * Unscheduled cardiac surgery anytime between enrollment to completion of the study.
  * Intra-procedure stroke
  * Radiation exposure ≥ 8 Gy
Freedom from major adverse event(MAE) | 30 days post-procedure
  Freedom from major adverse event(MAE) is defined as the freedom from device related MAE assessed through 30 days post-index procedure, as assessed by the Clinical Events Committee(CEC).

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, China